CLINICAL TRIAL: NCT06516718
Title: Post-marketing Observational Clinical Study: Assessment of the Effectiveness (Efficacy) of Odeston (Odeston®) in Patients With Chronic Cholecystitis in Real Medical Practice
Brief Title: An Assessment of the Effectiveness (Efficacy) of Odeston (Odeston®) in Patients With Chronic Cholecystitis in Real Medical Practice
Status: Not yet recruiting | Type: Observational
Sponsor: Kazakhstan Scientific Society for Study of intestine diseases (Other)
Responsible Party: Sponsor
Other Study IDs: UO-KSSSID-01
Record Dates: First submitted 2024-07-09; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Chronic Cholecystitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-marketing Observational Clinical Study: Assessment of the Effectiveness (Efficacy) of Odeston (Odeston®) in Patients With Chronic Cholecystitis in Real Medical Practice

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 65 years;
* BMI 18.5 - 40;
* Verified diagnosis: chronic acalculous cholecystitis;
* Voluntary desire to provide informed consent to participate in the study

Exclusion Criteria:

* Presence of stones in the gall bladder and bile ducts;
* The presence of jaundice, cholestatic liver diseases, liver cirrhosis with decompensation;
* Increased ALT, AST above the 3 upper limits of normal;
* Hypersensitivity to the components of the drug Odeston;
* Pregnancy and lactation;
* Prolonged fasting and total parenteral nutrition;
* Patients with symptoms of acute abdomen at the time of inclusion in the study;
* Patients with symptoms of acute neurological pathology at the time of inclusion in the study and/or аcute cerebrovascular accident, a history of convulsive syndrome;
* Presence of cancer;
* Acute infectious diseases at the time of inclusion in the study;
* Fever of any origin (above 37.5 C);
* Patients with symptoms of heart failure;
* Patients with symptoms of pulmonary failure;
* Patients with symptoms of acute or chronic renal failure;
* A decompensated form of diabetes;
* Patients with signs of psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes aged ≥18 to 65 years inclusive with a verified diagnosis: chronic acalculous cholecystitis
Sampling Method: Non-Probability Sample
Enrollment: 169 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Dynamics of Visual Analogue Scale scores for the severity and frequency of pain symptoms | on day 21

SECONDARY OUTCOMES:
Proportion of patients with a decrease in the severity of dyspeptic syndrome based on the Leeds Questionnaire | on day 21
Dynamics of quality of life indicators based on the Digestive Quality of Life Questionnaire | on day 21
Incidence of SUSAR | on day 21
The dynamics of Aspartate aminotransferase | on day 21
The dynamics of Alanine aminotransferase | on day 21
The dynamics of Alkaline phosphatase | on day 21
The dynamics of Gamma-glutamyl transpeptidase | on day 21
The dynamics of bilirubin with fractions | on day 21
Types of concomitant therapy uses | on day 21
Frequency of use of concomitant therapy | on day 21
Assessment of the shape of the gallbladder by ultrasound | on day 21
Assessment of the size of the gallbladder by ultrasound | on day 21
Assessment of the thickness of the gallbladder walls by ultrasound | on day 21
Assessment of the presence of intraluminal formations of the bladder by ultrasound | on day 21
Assessment of the presence of an acoustic shadow by ultrasound | on day 21
Assessment of the mobility of intraluminal formations by ultrasound | on day 21
Assessment of the presence of biliary sludge by ultrasound | on day 21
Assessment of the size of the common bile duct by ultrasound | on day 21
Assessment of the presence of dilatation of the intrahepatic bile ducts by ultrasound | on day 21
Assessment of the presence of additional formations using ultrasound | on day 21

CONTACTS AND LOCATIONS:
Locations (15):
- Kazakhstan (15):
  - "Human Health Clinic" LLP, Almaty
  - JSC "Research institute of cardiology and internal disease", Almaty
  - State-owned public enterprise with the right of economic management City Clinic No. 5, Almaty
  - "Taimas Medical" LLP, Astana
  - Medical center "Aiya", Astana
  - Medical Center Hospital of the President's affairs Administration of the Republic of Kazakhstan, Astana
  - NpJSC "Astana Medical University", Astana
  - State-owned public enterprise with the right of economic management "Multidisciplinary regional hospital" of the Kyzylorda Region Health Department, Kyzylorda
  - "Treatment Center No. 14" LLP, Shymkent
  - City diagnostic center of Shymkent, Shymkent
  - Medical Center "Aesculapius Vita", Shymkent
  - State-owned public enterprise with the right of economic management "District polyclinic Sauran" of the Department of Public Health of the Turkestan region, Shymkent
  - "Comec Medical Company" Llp, Taraz
  - "Hayat Medical Group" LLP Diagnostic Center, Taraz
  - Medical Center "Meyirim", Taraz